CLINICAL TRIAL: NCT00952939
Title: Prognostication of Uveal Melanoma by Fine Needle Aspiration (FNA) and Fluorescence in Situ Hybridization (FlSH)
Brief Title: Study of Tumor Samples in Patients Undergoing Radiation Therapy or Surgery For Primary Melanoma of the Eye
Status: Completed | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CASE5608; P30CA043703 (NIH); CASE5608 (Other: Case Comprehensive Cancer Center); CASE 5608-CC666 (Other: Cancer Center IRB)
Record Dates: First submitted 2009-08-05; First posted 2009-08-06 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Intraocular Melanoma
Keywords: ciliary body and choroid melanoma, small size; iris melanoma; intraocular melanoma; ciliary body and choroid melanoma, medium/large size
MeSH Terms: conditions — Uveal Melanoma | interventions — In Situ Hybridization, Fluorescence; Biopsy, Fine-Needle; Surveys and Questionnaires; 4-amino-4'-hydroxylaminodiphenylsulfone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: fluorescence in situ hybridization — At time of surgery
Other: laboratory biomarker analysis — At time of surgery
Procedure: fine-needle aspiration — At time of surgery
Procedure: therapeutic conventional surgery — At time of surgery
Other: Questionnaires — The MINI (a structured psychiatric interview) will be administered to all patients that had a pre or post-operative HADS score for suggestive or probable depression or anxiety. A semi-structured interview would be administered to those patients who had some or full decision regret pre-operatively. After completion of the interview, the MINI, a structured psychiatric interview, will be administered.
  Other Names: Hospital Anxiety and Depression Scale (HADS); Decision Regret Scale; The MINI (a structured psychiatric interview)

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This clinical trial is studying tumor samples in patients undergoing surgery or radiation therapy for primary melanoma of the eye.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To establish the feasibility of using fine needle aspiration (FNA) and FISH to determine tumor genotype in patients with primary uveal melanoma.

Secondary

* To characterize ophthalmic complication rate of FNA for FISH analysis in patients undergoing plaque radiotherapy.
* To estimate disease-free survival in patients with and without tumor monosomy 3 and/or 8q amplification.
* To explore the relationship between tumor monosomy 3 and 8q amplification and plasma levels of tumor immune escape and invasion biomarkers (e.g., circulating granulysin, beta2-microglobulin, autotoxin, lysophosphatidic acid, matrix metalloproteinase-7, tissue inhibitor of matrix metalloproteinase, and soluble E- cadherin).
* To explore the psychological impact of prognostication in uveal melanoma.

OUTLINE: Patients undergo plaque radiotherapy, enucleation, or tumor resection based upon standard of care guidelines.

Trans-scleral fine needle aspiration (FNA) is performed at the time of plaque radiotherapy and ex vivo FNA is performed on enucleation and tumor resection specimens. Tissue samples are analyzed by fluorescence in situ hybridization (FISH). Blood samples are also collected for further analysis.

After completion of study therapy, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria

* Patients must have a clinical diagnosis of melanoma of the iris, ciliary body and/or choroids
* Patients must have had a hepatic ultrasound and/or other suitable imaging studies to eliminate metastatic disease
* Patients must not have received any local or systemic therapy for uveal melanoma
* All patients must be informed of the investigational nature of this study and must provide written informed consent in accordance with institutional and federal guidelines. A copy of the informed consent document signed by the patient must be given to the patient
* Patients must have the following pretreatment laboratory findings:

  * Bilirubin (total) </= 1.5 ml/dl
  * AST </= 2 x normal
  * ALT </= 2 x normal
  * Alkaline phosphatase </= 2 x normal

Exclusion Criteria

* Patients with metastasis
* Patients under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2009-03; Primary Completion 2012-09 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Number of patients that have Disease Free Survival (DFS) with primary uveal melanoma with and without high-risk genotypes | 2 years
  DFS will be measured from the date of initial treatment to the date of documented recurrence or death. It will be summarized using the method of Kaplan and Meier.

SECONDARY OUTCOMES:
Number of patients with adverse events to determine ophthalmic complication rate of FNA for FISH analysis in patients undergoing plaque radiotherapy. | 2 years
  To characterize ophthalmic complication rate of FNA for FISH analysis in patients undergoing plaque radiotherapy.
The rate that sufficient tissue can be obtained by FNA. | 2 yrs
  Determine if sufficient material for FISH analysis can be obtained by transscleral FNA, a diagnostic procedure performed for a variety of clinical indications in patients with eye abnormalities.
distribution of particular markers at specific timepoints | at baseline, multiple time points up to 2 years
  Plasma will be analyzed for circulating granulysin, beta2-microglobulin, autotoxin, lysophosphatidic acid, matrix metalloproteinase-7, tissue inhibitor of matrix metalloproteinase, and soluble E-cadherin.

CONTACTS AND LOCATIONS:
Overall Officials: Arun D. Singh, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Cole Eye Institute, Cleveland, Ohio, United States